CLINICAL TRIAL: NCT00970086
Title: Transversus Abdominis Plane Block for Pain Relieve in Children Undergoing Inguinal Surgical Procedures: How Does it Compare With the "Gold Standard" Caudal Blockade
Brief Title: Transversus Abdominis Plane Block for Pain Relieve in Children Undergoing Groin Surgery
Acronym: TAP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Groin surgery was changed to a laparoscopic technique; recruitable patients ceased.
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: UKBB_ANA_TAP
Record Dates: First submitted 2009-08-25; First posted 2009-09-02 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Postoperative Pain; Reaction; Anesthesia
Keywords: measure of postoperative pain; children undergoing groin surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- transversus abdominal plane block (Experimental): Caudal block: Identification of the epidural space with a loss of resistance technique. Administration of Bupivacain 1ml/kg 0.125%.
  Transversus abdominal plane block: Identification of the anatomical structures with ultrasound, insertion of the stimuplex needle G22, 50mm, in an in-plane approach and administration of 0.4ml/kg levobupivacaine 0.25%.
  Interventions: Drug: Bupivacain/levobupivacaine

INTERVENTIONS:
Drug: Bupivacain/levobupivacaine — Caudal block: Identification of the epidural space with a loss of resistance technique. Administration of Bupivacain 1ml/kg 0.125%.
  Transversus abdominal plane block: Identification of the anatomical structures by the ultrasound technique, administration of 0.4ml/kg levobupivacaine 0.25%.

SUMMARY:
For surgery in the region of the lower abdominal wall the administration of local anesthetic drugs in the epidural space via the caudal route is the preferentially used technique since several decades.

The transversus abdominis plane (TAP) block features the advantages of a peripheral nerve blockade. The aim of this study is to evaluate potential differences in the effectiveness of postoperative analgesia and to test the hypotheses that the duration of pain relieve ist prolonged after a TAP block when compared with an epidural technique.

DETAILED DESCRIPTION:
Caudal block (CB) is the gold standard technique for analgesia in children undergoing surgical interventions in the groin.

Although the efficacy and the safety of this technique is high, nonetheless, there are several caveats such as unwarranted motor blockade of the lower limbs and disturbances of the bladder function, potentially resulting in delayed demission in the ambulatory setting. The effect of the blockade wears off within 4-5h post-block, making the administration of additional pain medication necessary.

Peripheral nerve blockades (PNB) are an alternative to CB and have a prolonged duration of the analgesic effect. More recently, an alternative method to block neural structures which innervate lower abdominal wall has been described; the transverse abdominal plane block. The ultrasound guided technique improves the safety of margin. However, although this new technique seems to offer substantial advantages so far only experience from small case series are available. In particular, the TAP block has not been compared in a systematic trial with the "gold standard", the caudal block.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children aged 2 - 8 years
* physical status classification system (ASA) score I or II
* Undergoing surgical interventions in the groin (hernia repair, funiculocele ectomy)

Exclusion Criteria:

* Hypersensitivity to Levobupivacaine

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2009-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of the postoperative analgesia: monitoring with KUSS or Smiley scale. | 4 h postoperative and morning, 1 day postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Erb, PD, Principal Investigator — University Childrens Hospital of both Basel
Locations (1):
- University Childrens Hospital of both Basel, Basel, Basel, Switzerland